CLINICAL TRIAL: NCT04174885
Title: Calcium Handling and SERCA Protein Activity Modulation in Patients With Persistent Atrial Fibrillation (AF) Treated by Epicardial Thoracoscopic Ablation: the CAMAF Study
Brief Title: Calcium Handling and Epicardial Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, principal investigator, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SecondUNI 18.11.2019
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AF epicardial ablation (Other): Patient with persistent AF will receive an epicardial ablation.
  Interventions: Procedure: epicardial ablation

INTERVENTIONS:
Procedure: epicardial ablation — In general anesthesia and left lung ventilation, authors will access the right thorax by three working ports. However, a rigid video thoracoscopic camera with a direct optics will be used. Pericardium will be widely opened anterior to a phrenic nerve and transverse and oblique sinuses were dissected. An insertion of the ablation catheter will be a tricky part of the surgery with the first MW catheter, while no special introducer will be provided. Later RF devices will be equipped with a special flexible introducers, lately also with a magnetic tip and the positioning of the catheter around PVs became much safer and easier.
  The correct position of catheter will be visualized by trans esophageal echocardiography before the ablation.

SUMMARY:
In this multi centre prospective study authors will evaluate atrial fibrillation (AF) recurrence at 360 days follow-up and calcium handling in patients treated by epicardial thoracoscopic ablation for persistent AF. Indeed, responders patients to epicardial ablation will experience sinus rhythm restoration after the treatment, and will be in sinus rhythm until follow-up end.

However, from October 2014 to June 2016, 27 consecutive patients with persistent AF will be identified and screened for participation in this prospective, multicenter trial at Catholic University of Sacred Heart, Campobasso, at University Study of Molise, Campobasso, at Vecchio Pellegrini Hospital, Naples and at University of Campania "Luigi Vanvitelli", Naples, Italy. All patients will receive an epicardial thoracoscopic pulmonary vein isolation. Before interventions, baseline laboratory studies, B type Natriuretic Peptide (BNP) and serum Sarcoplasmic Endoplasmic Reticulum Calcium ATPase (SERCA) will be evaluated. These markers will be re-evaluated at 12th month of follow-up.

Therefore, study hypothesis will be that successful epicardial ablation might reduce, in responders patients, the SERCA expression. Parallely, a lower serum expression of SERCA in patients with persistent AF might potentially identify a response to an epicardial ablative approach, and an innovative target to improve the response to an epicardial ablative treatment.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is most common arrhythmia in the worldwide population, and it is defined as paroxysmal, persistent and/or permanent. Patients with persistent AF might have higher rate of tromboembolic stroke, heart failure events and worse prognosis. Therefore, for patients with persistent AF the sinus rhythm restoration by catheter ablation might be a valid treatment to ameliorate clinical outcomes. On other hand, in patients with persistent AF the catheter ablation by percutaneous approach has a success rate about the 50% at 5 years of follow-up. Indeed, the endocardial ablation cannot determine deeper and extensive trans mural lesions in pulmonary veins and left atrium structure, and this might favor atrial fibrosis and remodeling with consequent persistence of arrhythmic substrate. In this setting, the epicardial AF ablation has been proposed to reach epicardial gaps of the complex arrhythmic atrial substrate, and this might favor sinus rhythm restoration with consequent reduction of the left atrial diameters and volume in patients with persistent AF. Notably, 40% of patients treated by epicardial ablatiion might show an AF recurrence at follow-up. This might be explained by multiple ionic, molecular and cellular alterations favoring AF persistence. In this setting, recently a great interest has been focused to study the calcium handling as cause of abnormal trigger activity and reentry in AF patients, that are both mechanisms implied in the genesis and perpetuation of persistent AF. Intriguingly, patients with persistent AF have an over activity of the Sarcoplasmic Endoplasmic Reticulum (SR) with increased calcium (Ca2+) release. However, in human atrial myocites the Ca2+ overload causes an increased prevalence of spontaneous events and delayed after depolarizations (DADs), (12). Therefore, the SERCA over activity increases the risk of Ca overload and this might be arrhythmogenic (13). Therefore, abnormal Ca2+ signaling and enhanced diastolic SR Ca2+ leak along with cellular DAD-mediated triggered activity might promote AF persistence, than favoring electrical and anatomical reentry. Conversely, the persistence of abnormal Ca2+ signaling and enhanced diastolic SR Ca2+ leak can activate ion channels and trigger Ca2+-dependent signaling pathways, thereby promoting the evolution of atrial remodeling and the progression of AF to more persistent forms. In this setting, authors might speculate that these AF-related alterations in Ca2+ handling and SERCA over activity might contribute to AF persistence after an epicardial ablation. Intriguingly, no data have been reported about the SERCA activity in patients with persistent AF before and after epicardial ablation. Moreover, authors study hypothesis is that a SERCA over expression might be linked to higher rate of failure to an epicardial ablation for patients with persistent AF. Thereafter, in this study authors will evaluate AF recurrences during 1 year of follow-up after epicardial ablation, correlating this clinical outcomes to SERCA protein modifications in patients with sinus rhythm restoration (responders group), vs. atrial fibrillating patients (non responders group) after an epicardial ablative approach.

ELIGIBILITY:
Inclusion Criteria:

* persistent AF, both genders, aged >18 years, aged < 75 years.

Exclusion Criteria:

* neoplastic diseases, inflammatory chronic diseases, acute and chronic heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence. | 12 months
  Authors will evaluate the atrial fibrillation recurrence at 12 months of follow-up after epicardial ablation. Atrial fibrillation recurrence will be measured during clinical visits, and by the registration of 12 derivations electrogram (ECG), and ECG Holter.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Celestino Sardu, Naples
  - Raffaele Marfella, Naples

IPD SHARING:
Plan to Share IPD: Undecided